CLINICAL TRIAL: NCT05666219
Title: Assessing the Impact of Aminophylline in the Reversal of Complete Heart Block Secondary to Inferior Wall MI in Atropine Resistant Patients: An Open Label Non-randomized Clinical Trial
Brief Title: Reversal of Complete Heart Block With Aminophylline in Inferior Wall Myocardial Infarction Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: we could not find patients fulfilling all of our inclusion criteria
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC-32/2022
Record Dates: First submitted 2022-12-13; First posted 2022-12-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Complete Heart Block; Inferior Wall Myocardial Infarction
MeSH Terms: conditions — Inferior Wall Myocardial Infarction | interventions — Aminophylline; Theophylline

STUDY DESIGN:
Intervention Model Description: An Open Label Non-randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment group (Experimental): Patients receiving Injection Aminophylline
  Interventions: Drug: Aminophylline Injection

INTERVENTIONS:
Drug: Aminophylline Injection — Injection Aminophylline IV 240 mg will be given over 10 minutes. After 1 hour, Aminophylline 240 mg second dose will be given over 10 minutes.
  Other Names: Theophylline

SUMMARY:
In this study, the investigator will evaluate the rate of reversal of complete heart block with aminophylline in atropine resistant patients with inferior wall myocardial infarction (MI)

DETAILED DESCRIPTION:
Administration of Aminophylline can result in reversal of complete heart block in a significant number of atropine resistant patients with inferior wall MI. Hence, in this study our primary aim is to evaluate the rate of reversal of complete heart block with aminophylline in atropine resistant patients with inferior wall MI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted with recent acute inferior wall myocardial infarction (MI)
* Hemodynamically stable blood pressure
* Complete heart block with Narrow QRS < 120 ms and ventricular rate >40/min persisting for at least 6 hours, resistant to atropine
* Temporary pacemaker (TPM) already placed
* Patient asymptomatic with a mean arterial pressure of greater than 65 mmHg with TPM rate placed at 40/min

Exclusion Criteria:

* Patients with cardiogenic shock
* Patients with preexisting permanent pacemaker and Implantable Cardioverter Defibrillator (ICD).
* Patients with a prior history of AV block
* Drugs with dromotropic effects (beta blocker, calcium channel blocker, inotropes)
* Known liver disease (cirrhosis, hepatitis)
* Hypothyroidism
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Reversal of complete heart block | Within 1 hour of 2nd dose
  Conversion to sinus rhythm with 1:1 conduction

SECONDARY OUTCOMES:
Improved conduction | Within 1 hour of 2nd dose
  Combined end point of 1:1 conduction and improved conduction to second degree AV block
Major adverse cardiac events (MACE) | Within 12 hours
  Ventricular arrhythmias ( VT more than 3 beats), decrease in ventricular escape rate requiring increasing pacing rate, cardiac arrest or death

CONTACTS AND LOCATIONS:
Overall Officials: Azam Shafquat, MD, Study Chair — National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
No individual participant data sharing plan in placed